CLINICAL TRIAL: NCT04754373
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Study to Evaluate the Effect of GFA-918 on Serum Triglyceride Levels in Individuals With Elevated Serum Triglyceride
Brief Title: A Study to Evaluate the Effect of GFA-918 on Serum Triglyceride Levels in Individuals With Elevated Serum Triglyceride
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BIO-CAT Microbials, LLC (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Organization: BIO-CAT, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 17GTHB
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-10

CONDITIONS: Elevated Triglycerides
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GFA-918 (Experimental): Participants will be instructed to take one GFA-918 capsule twice per day with their morning and evening meals for 12 weeks.
  Interventions: Dietary Supplement: GFA-918
- Placebo (Placebo Comparator): Participants will be instructed to take one Placebo capsule twice per day with their morning and evening meals for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: GFA-918 — Participants will be instructed to take one GFA-918 (125000 FIP Units of Lipase AY) capsule twice per day with their morning and evening meals for 12 weeks.
  Arms: GFA-918
Other: Placebo — Participants will be instructed to take one Placebo capsule twice per day with their morning and evening meals for 12 weeks.
  Arms: Placebo

SUMMARY:
In this study, a lipase -sourced from a nonpyrogenic yeast, Candida rugosa, will be investigated to establish optimal TG levels in adults in a 12-week supplementation period. The investigational product provides a lipase formulation that is stable and active in acidic and neutral pH environments, while also fully digesting TGs into free fatty acids and glycerol which is beyond the scope of pancreatic lipase (Schuler et al. 2012). This will be a novel study investigating the effects of C. rugosa lipase on adults with slightly elevated TG levels.

ELIGIBILITY:
Inclusion Criteria:

1. Females and male within the age range of 30 to 70 at screening;
2. BMI of 20 - 34.9 kg/m2 at screening;
3. Not of child bearing potential, which is defined as females who have had hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation) OR,

   Female participants of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result, prior to enrollment. All hormonal birth controls require a minimum stability of three months and remain consistent throughout the study. Acceptable methods of birth control include:
   * Hormonal contraceptives; oral, hormone patch (Ortho Evra), vaginal ring (NuvaRing), injectable (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner (shown successful as per appropriate follow-up);
4. Sedentary life style as defined by Sedentary Behavior Questionnaire (Appendix II) at screening;
5. Serum triglycerides 1.91 - 3.93 mmol/L (175 - 350 mg/dL) (inclusive) at screening;
6. Willing to maintain current levels of activity throughout the study;
7. Stable with no health concerns for participating in the study as determined by laboratory results, and medical history;
8. Willingness to complete all study visits and requirements associated with the study;
9. Has access to a computer, tablet, or smart phone with internet connection;
10. Has given voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

1. Individuals who are pregnant, breastfeeding, or planning to become pregnant;
2. LDL-C ≥ 4.1 mmol/L (160 mg/dL);
3. Uncontrolled hypertension, defined as untreated systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 90 mmHg;
4. Cancer(s), except skin cancers completely excised with no chemotherapy or radiation with a negative follow up. and cancer(s) in full remission for more than five years after diagnosis
5. Immunocompromised individuals such as those that have undergone organ transplantation, those with rheumatoid arthritis, or those diagnosed with human immunodeficiency virus (HIV) or AIDS by verbal confirmation;
6. Verbal confirmation of current, or history of, bleeding disorders and/or medically prescribed anticoagulant/antiplatelet drugs (refer to Section 5.3);
7. Verbal confirmation of current unstable thyroid disease state; however, participants who have been on stable medication for >6 months will be eligible to participate but will be assessed on a case by case basis by the QI.
8. Verbal confirmation of GI disorders and on anti-inflammatory drugs to control GI disorders; however, participants who have been on stable medication for >6 months will be eligible to participate but will be assessed on a case by case basis by the QI
9. Verbal confirmation of Type I and Type II Diabetes;
10. Anti-inflammatory medication, corticosteroids, lipid lowering agents and diabetic medication (refer to Section 5.3) as assessed by the QI;
11. Alcohol or drug abuse within the last 6 months;
12. No more than 2 standard alcoholic drinks per day;
13. Verbal confirmation of marijuana use >4 times a week
14. Tobacco products, including e-cigarette; dose and frequency will be assessed on a case by case basis by the QI
15. Participation in a clinical research study within 30 days of enrollment;
16. Allergy or sensitivity to study product ingredients;
17. Clinically significant abnormal laboratory results at screening;
18. Unstable medical conditions as assessed by the Qualified Investigator;
19. Individuals who are cognitively impaired and/or unable to give informed consent;
20. Any other condition which in the Qualified Investigator's opinion may adversely affect the participant's ability to complete the study or its measures or which may pose significant risk to the participant.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
The change in levels of fasting serum TG levels | 12 weeks
  The primary outcome of this study is the change in levels of fasting serum TG levels from screening to week 12 in fasting serum TG levels between GFA-918 and placebo groups.

SECONDARY OUTCOMES:
The change in levels of triglycerides | 12 weeks
  The change from baseline to week 12 in lipid profile (levels of triglycerides) between GFA-918 and placebo groups
The change in levels of total cholesterol | 12 weeks
  The change from baseline to week 12 in lipid profile (levels of total cholesterol) between GFA-918 and placebo groups
The change in levels of LDL-cholesterol | 12 weeks
  The change from baseline to week 12 in lipid profile ( levels of LDL-cholesterol) between GFA-918 and placebo groups
The change in levels of VLDL-cholesterol | 12 weeks
  The change from baseline to week 12 in lipid profile (levels of VLDL-cholesterol) between GFA-918 and placebo groups
The change in levels of HDL-cholesterol | 12 weeks
  The change from baseline to week 12 in lipid profile (levels of HDL-cholesterol) between GFA-918 and placebo groups
The change in levels of ApoA-I | 12 weeks
  The change from baseline to week 12 in lipid profile (levels of ApoA-I) between GFA-918 and placebo groups
The change in levels of LDL-C: HDL-C | 12 weeks
  The change from baseline to week 12 in lipid profile (LDL-C: HDL-C) between GFA-918 and placebo groups
The change in levels of TC: HDL-C | 12 weeks
  The change from baseline to week 12 in lipid profile (TC: HDL-C) between GFA-918 and placebo groups
The change in levels of apolipoprotein A1 (ApoA-1) | 12 weeks
  The change from baseline to week 12 in apolipoprotein A1 (levels of ApoA-1) between GFA-918 and placebo groups.
The change in levels of CRP | 12 weeks
  The change from baseline to week 12 in levels of the inflammatory biomarker, CRP, between the GFA-918 and placebo groups
The change in levels of TNF-α | 12 weeks
  The change from baseline to week 12 in levels of the inflammatory biomarker, TNF-α, between the GFA-918 and placebo groups
The change in levels of IL-6 | 12 weeks
  The change from baseline to week 12 in levels of the inflammatory biomarker, IL-6, between the GFA-918 and placebo groups
The change in body weight | 12 weeks
  The change from screening to week 12 in body weight between GFA-918 and placebo groups.
The change in body mass index (BMI) | 12 weeks
  The change from screening to week 12 in body mass index (BMI) between the GFA-918 and placebo groups
A clinically relevant change in TG after the 12-week supplementation with GFA-918 as assessed by a 1 mmol/L decrease in TG. | 12 weeks
  6A clinically relevant change in TG from screening to week 12 after the 12-week supplementation with GFA-918 as assessed by a 1 mmol/L decrease in TG.
A clinically relevant change in HDL-C after supplementation with GFA-918 defined as at least 0.026 mmol/L (1 mg/dL) or 1% increase | 12 weeks
  A clinically relevant change in HDL-C, from baseline to week 12 after supplementation with GFA-918 defined as at least 0.026 mmol/L (1 mg/dL) or 1% increase
The clinically relevant change in LDL-C after supplementation with GFA-918 defined as a minimal 1% decrease | 12 weeks
  The clinically relevant change in LDL-C, from baseline to week 12 after supplementation with GFA-918 defined as a minimal 1% decrease
The changes during the follow up period, week 12 to week 14, in levels of fasting serum TG levels | 14 weeks
  The changes during the follow up period, week 12 to week 14, in fasting serum TG levels between GFA-918 and placebo groups.
The changes during the follow up period, week 12 to week 14, in complete lipid profile | 14 weeks
  The changes during the follow up period, week 12 to week 14, complete lipid profile between GFA-918 and placebo groups.
The changes during the follow up period, week 12 to week 14, in levels of ApoA-1 | 14 weeks
  The changes during the follow up period, week 12 to week 14, ApoA-1, between GFA-918 and placebo groups.
The changes during the follow up period, week 12 to week 14, in levels of inflammatory biomarkers | 14 weeks
  The changes during the follow up period, week 12 to week 14, inflammatory biomarkers, between GFA-918 and placebo groups.
The changes during the follow up period, week 12 to week 14, in body weight | 14 weeks
  The changes during the follow up period, week 12 to week 14, body weight between GFA-918 and placebo groups.
The changes during the follow up period, week 12 to week 14, in BMI | 14 weeks
  The changes during the follow up period, week 12 to week 14, BMI, between GFA-918 and placebo groups.
The clinical significant changes during the follow up period, week 12 to week 14, in levels of TG | 14 weeks
  The clinical significant changes during the follow up period, week 12 to week 14, in TG, between GFA-918 and placebo groups.
The clinical significant changes during the follow up period, week 12 to week 14, in levels of HDL-C | 14 weeks
  The clinical significant changes during the follow up period, week 12 to week 14, in HDL-C, between GFA-918 and placebo groups.
The clinical significant changes during the follow up period, week 12 to week 14, in levels of LDL-C | 14 weeks
  The clinical significant changes during the follow up period, week 12 to week 14, in LDL-C, between GFA-918 and placebo groups.

OTHER OUTCOMES:
The incidence of adverse events with GFA-918. | 12 weeks
  The incidence of adverse events during the 12-week supplementation with GFA-918.
The incidence of any abnormal vital signs: blood pressure (BP) and heart rate (HR), with GFA-918 | 12 weeks
  The incidence of any abnormal vital signs: blood pressure (BP) and heart rate (HR), during the 12-week supplementation with GFA-918
The incidence of any abnormal ECG with GFA-918 | 12 weeks
  The incidence of any abnormal ECG during the 12-week supplementation with GFA-918
The incidence of any abnormal hematology (white blood cell (WBC) count with differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils) with GFA-918. | 12 weeks
  The incidence of any abnormal hematology; white blood cell (WBC) count with differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils; during the 12-week supplementation with GFA-918.
The incidence of any abnormal hematology; red blood cell (RBC) count, with GFA-918. | 12 weeks
  The incidence of any abnormal hematology; hemoglobin, during the 12-week supplementation with GFA-918.
The incidence of any abnormal hematology; hematocrit, with GFA-918. | 12 weeks
  The incidence of any abnormal hematology; hematocrit, during the 12-week supplementation with GFA-918.
The incidence of any abnormal hematology; platelet count, with GFA-918. | 12 weeks
  The incidence of any abnormal hematology; platelet count, during the 12-week supplementation with GFA-918.
The incidence of any abnormal hematology; RBC indices (mean corpuscular volume (MCV)) with GFA-918. | 12 weeks
  The incidence of any abnormal hematology; RBC indices (mean corpuscular volume (MCV)), during the 12-week supplementation with GFA-918.
The incidence of any abnormal hematology; RBC indices (mean corpuscular hemoglobin (MCH)), with GFA-918. | 12 weeks
  The incidence of any abnormal hematology; RBC indices (mean corpuscular hemoglobin (MCH), during the 12-week supplementation with GFA-918.
The incidence of any abnormal hematology; RBC indices (mean corpuscular hemoglobin concentration (MCHC)), with GFA-918. | 12 weeks
  The incidence of any abnormal hematology; RBC indices (mean corpuscular hemoglobin concentration (MCHC)) during the 12-week supplementation with GFA-918.
The incidence of any abnormal hematology; RBC indices (red cell distribution width (RDW)) with GFA-918. | 12 weeks
  The incidence of any abnormal hematology; RBC indices (red cell distribution width (RDW)) during the 12-week supplementation with GFA-918.
The incidence of any abnormal liver function measured: alanine aminotransferase (ALT), with GFA-918. | 12 weeks
  The incidence of any abnormal liver function measured: alanine aminotransferase (ALT), during the 12-week supplementation with GFA-918.
The incidence of any abnormal liver function measured: aspartate aminotransferase (AST), with GFA-918. | 12 weeks
  The incidence of any abnormal liver function measured: aspartate aminotransferase (AST), during the 12-week supplementation with GFA-918.
The incidence of any abnormal liver function measured: bilirubin, with GFA-918. | 12 weeks
  The incidence of any abnormal liver function measured: bilirubin, during the 12-week supplementation with GFA-918.
The incidence of any abnormal kidney function parameters: serum creatinine, with GFA-918 | 12 weeks
  The incidence of any abnormal kidney function parameters: serum creatinine, during the 12-week supplementation with GFA-918
The incidence of any abnormal kidney function parameters: estimated glomerular filtration rate (eGFR), with GFA-918 | 12 weeks
  The incidence of any abnormal kidney function parameters: estimated glomerular filtration rate (eGFR), during the 12-week supplementation with GFA-918
The incidence of any abnormal kidney function parameters: electrolytes (Na, K, Cl), with GFA-918 | 12 weeks
  The incidence of any abnormal kidney function parameters: electrolytes (Na, K, Cl), during the 12-week supplementation with GFA-918
The incidence of any abnormal urinalysis measurements: colour | 12 weeks
  The incidence of any abnormal urinalysis measurements: colour, during the 12-week supplementation with GFA-918.
The incidence of any abnormal urinalysis measurements: appearance | 12 weeks
  The incidence of any abnormal urinalysis measurements: appearance, during the 12-week supplementation with GFA-918.
The incidence of any abnormal urinalysis measurements: specific gravity | 12 weeks
  The incidence of any abnormal urinalysis measurements: specific gravity, during the 12-week supplementation with GFA-918.
The incidence of any abnormal urinalysis measurements: pH | 12 weeks
  The incidence of any abnormal urinalysis measurements: pH, during the 12-week supplementation with GFA-918.
The incidence of any abnormal urinalysis measurements: presence of protein | 12 weeks
  The incidence of any abnormal urinalysis measurements: presence of protein, during the 12-week supplementation with GFA-918.
The incidence of any abnormal urinalysis measurements: glucose | 12 weeks
  The incidence of any abnormal urinalysis measurements: glucose, during the 12-week supplementation with GFA-918.
The incidence of any abnormal urinalysis measurements: ketones | 12 weeks
  The incidence of any abnormal urinalysis measurements: ketones, during the 12-week supplementation with GFA-918.
The incidence of any abnormal urinalysis measurements: blood | 12 weeks
  The incidence of any abnormal urinalysis measurements: blood, during the 12-week supplementation with GFA-918.
The incidence of any abnormal urinalysis measurements: nitrites | 12 weeks
  The incidence of any abnormal urinalysis measurements: nitrites, during the 12-week supplementation with GFA-918.
The incidence of any abnormal urinalysis measurements: leucocyte esterase | 12 weeks
  The incidence of any abnormal urinalysis measurements: leucocyte esterase, during the 12-week supplementation with GFA-918.
The incidence of adverse events or abnormal safety outcomes during the follow up period, week 12 to week 14 | 14 weeks
  The incidence of adverse events or abnormal safety outcomes during the follow up period, week 12 to week 14

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science
Locations (2):
- Canada (2):
  - KGK Science, London, Ontario
  - Canadian College of Naturopathic Medicine, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No